CLINICAL TRIAL: NCT04654377
Title: Impact of Personalized Education on Pain Response in Patients With Chronic Pancreatitis (PEPCP)
Brief Title: Personalized Education and Pain Response in Chronic Pancreatitis
Acronym: PEPCP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Rupjyoti Talukdar, Director, Pancreatology; Head, Pancreas Research Group and Division of Gut Microbiome Research, Asian Institute of Gastroenterology, India
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PEPCP2023 ver 04
Record Dates: First submitted 2020-11-27; First posted 2020-12-04 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Chronic Pancreatitis; Pain Syndrome; Depression, Anxiety
Keywords: chronic pancreatitis; pain; depression; anxiety; quality of life; metabolome; magnetic resonance spectroscopy; quantitative sensory testing
MeSH Terms: conditions — Pancreatitis, Chronic; Somatoform Disorders; Depression; Anxiety Disorders; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Personalised education (Experimental): 1. Greetings.
  2. Recording of demographic, clinical (disease related), nutritional, laboratory, and treatment related data.
  3. Administration of questionnaires.
  4. Inquiring patient's perception of their disease.
  5. Explaining the patient about their disease in general followed by specific aspects and possible outcomes in the context of their perception, clinical aspects, questionnaire, and imaging data. In addition, the general treatment plan will be explained.
  6. Address all queries from the patient and care givers.
  Interventions: Other: Personalised education
- Standard communication (No Intervention): 1. Greetings.
  2. Recording of demographic, clinical (disease related), nutritional, laboratory, imaging and treatment related data.
  3. Administration of questionnaires.
  4. Explaining the general treatment plan.
  5. Address general treatment related queries from the patient and care givers.

INTERVENTIONS:
Other: Personalised education — Patients will be explained about their disease and possible outcomes based on clinical, biochemical and imaging data.
  Arms: Personalised education

SUMMARY:
Pain mechanisms in chronic pancreatitis (CP) are heterogeneous and includes nociception, pancreatic neuropathy and central neuropathy/neuroplasty. These mechanisms could occur simultaneously in variable proportions and could explain why several patients develop recurrence of pain even after being treated by all the currently available modalities, such as antioxidants, endoscopic therapies and surgery.

In the studies by the investigators over the past 2 years, they observed that persistent pain in these patients was associated with varying grades of depression and poor quality of life. This was accompanied by alteration in the metabolites in the brain (anterior cingulate cortex, prefrontal cortex, hippocampus, and basal ganglia) as evidenced in magnetic resonance spectroscopy (MRS) of the brain. These areas in the brain are responsible for pain modulation, long-term pain memory and emotional responses to pain.

When the investigators counselled these patients and explained their disease and possible outcomes based on their own clinical course, imaging and treatment response (personalized education/counselling), they reported significant improvement in depression, quality of life parameters and, interestingly, also in pain. Further, there were changes in the metabolite parameters in the brain on MRS after personalized counselling/education that was more similar to that of healthy controls.

This led to our hypothesis that better understanding of the disease and its outcomes by the patients could improve their coping capabilities and increase their pain thresholds. This could augment the pain responses of these patients to the other therapeutic modalities.

We will conduct this single blinded, placebo controlled, randomized controlled trial on patients with documented CP of over 3 years duration, who had at least 3 episodes of abdominal pain of over the past 3 months.

DETAILED DESCRIPTION:
Chronic pancreatitis (CP) is characterised by pain, exocrine insufficiency and endocrine dysfunction. Of all symptoms, intractable abdominal pain is the most debilitating that mandates a multidisciplinary treatment approach. Long term treatment of pain begins with antioxidants. If the pancreatic duct contains stones in a limited area (head, neck and proximal body), the patient is subjected to endoscopic treatment, which includes extracorporeal shock wave lithotripsy (ESWL) for large stones (>5mm) with or without pancreatic duct stenting. For smaller stones, endoscopic retrograde cholangiopancreatography (ERCP) alone suffices. ERCP with pancreatic ductal stenting is also the first line treatment for a solitary symptomatic pancreatic ductal stricture. If symptomatic stones are located all along the pancreatic duct, or if there are multiple strictures, surgical drainage of the pancreatic duct becomes the treatment of choice. If there are any mass lesion in the pancreas on the background of CP, then resection procedures such as Whipple's operation or distal pancreatectomy with/without splenectomy is resorted to.

Even though the above mentioned modalities are directed to relief the patient of pain, a substantial proportion of patients return with recurrence of pain. This explains the complexity in the pain mechanisms in CP. Pain mechanisms in chronic pancreatitis (CP) are heterogeneous and includes nociception, pancreatic neuropathy and central neuropathy/neuroplasticity. These mechanisms could occur simultaneously in variable proportions and could explain why several patients develop recurrence of pain even after being treated by all the currently available modalities.

Since CP is a chronic disease with systemic effects, several additional factors could impact the evolution and response to pain. These could include the patient's personality traits, educational background, family history of CP, previous experience of the disease, background knowledge of CP, coping capability, to name a few. The investigators have been working on these aspects for the past couple of years, wherein they looked into the mental status (depression/anxiety), quality of life and the impact of pain in these aspects. Since pain memory and emotional responses to pain is mediated by the basal ganglia, hippocampus, anterior cingulate cortex and prefrontal cortex of the brain, the investigators also looked at the metabolites in these areas using magnetic resonance spectroscopy. The investigators observed that persistent pain in these patients will be associated with varying grades of depression and poor quality of life. This was accompanied by alteration in the metabolites myoinositol, creatine, glycine/glutamate in the hippocampus, and basal ganglia Following this, when the investigators counselled these patients and explained their disease and possible outcomes based on their own clinical course, imaging and treatment response (personalized education/counselling), they reported significant improvement in depression, quality of life parameters and, interestingly, also in pain. Further, there were changes in the metabolite parameters in the brain on MRS after personalized counselling/education that were more closer to that of healthy controls.

This led to the hypothesis that better understanding of the disease and its outcomes by the patients could improve their coping capabilities and increase their pain thresholds. This could augment the pain responses of these patients to the other therapeutic modalities.

The investigators will conduct this single blinded, placebo controlled, randomized controlled trial on patients with documented CP of over 3 years duration, who had at least 3 episodes of abdominal pain of over the past 3 months.

The investigators will provide detailed education regarding the disease to the patients (based on their disease characteristics) in the study arm and evaluate the changes in pain scores, pain episodes, QOL, mental status and metabolomic status in the brain (hippocampus, basal ganglia, anterior cingulate cortex, prefrontal cortex).

ELIGIBILITY:
Inclusion Criteria:

* Chronic pancreatitis of at least 3 years
* At least 3 episodes of pain in the past 3 months
* Age 18-60yrs
* Both genders

Exclusion Criteria:

* Acute pancreatitis episode at the time of enrolment.
* Pancreatic cancer.
* Other chronic diseases (including end organ damage related to diabetes).
* Adverse life event in the family in the past 6 months.
* Active substance use (alcohol, smoking, smokeless tobacco, Illicit drugs).
* Pregnancy and lactation.
* Psychiatric illness at enrolment or during follow-up, and/or concomitant intake of antidepressants and neuromodulators..

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 114 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in pain score | 3 and 6 months
  Pain will be measured using the Visual analog scale (0-10)

SECONDARY OUTCOMES:
Change in number of painful days | 3 and 6 months
  The patient will record the number of painful days in a self reported pain questionnaire.
Change in the number of hospital visits | 3 and 6 months
  The patient will record the number of hospital visits in a self reported daily questionnaire.
Change in neuropathic pain | 3 and 6 months
  Neuropathic pain will be evaluated using the PainDetect tool
Change in quality of life (QOL) | 3 and 6 months
  Quality of life (QOL) will be measured using the EORTC QLQ 30
Change in depression score | 3 and 6 months
  Depression will be measured using Beck depression Inventory (BDI) II
Change in depression score | 3 and 6 months
  Depression will be measured using Hospital Anxiety and Depression Score (HADS).
Change in anxiety score | 3 and 6 months
  Anxiety will be measured using the Hospital anxiety and depression (HADS) tools.
Change in multidimensional aspects of pain | 3 and 6 months
  Multidimensional aspects of pain will be measured using the COMPAT-SF
Change in the psychological aspects of pain | 3 and 6 months
  Psychological aspects of pain will be measured using the Pain Catastrophising score (PCS)
Change in sleep behaviour | 3 and 6 months
  Change in sleep behaviour will be measured using the Pittsburg Sleep Quality Index
Change in the patient's perception of alteration in pain | 3 and 6 months
  Patient's perception of alteration in pain will be measured using the Patient's Global Impression of Pain (PGIC)
Difference in analgesic requirement | 3 and 6 months
  Difference in analgesic requirement will be measured by number of opioids and NSAIDs requirement

OTHER OUTCOMES:
Evaluation of possible mechanisms of improvement. | 3 and 6 months
  Possible mechanisms of improvement improvement will be assessed by measuring the plasma metabolites serotonin, dopamine, oxytocin, GABA, tryptophan and endorphins.

CONTACTS AND LOCATIONS:
Overall Officials: Rupjyoti Talukdar, MD, FICP, AGAF, Principal Investigator — Asian Institute of Gastroenterology
Locations (1):
- Asian Institute of Gastroenterology, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: Yes
If other researchers collaborate with us in the future for similar research project, we will share de-identified data pertaining to patients clinical characteristics as per requirement of the study design.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After completion of study to one year thereafter.
Access Criteria: Collaborative study with similar study design/outcomes

REFERENCES:
- [Background] Talukdar R, Reddy DN. Pain in chronic pancreatitis: managing beyond the pancreatic duct. World J Gastroenterol. 2013 Oct 14;19(38):6319-28. doi: 10.3748/wjg.v19.i38.6319. PMID 24151350
- [Background] Talukdar R, Nageshwar Reddy D. Is there a single therapeutic target for chronic pancreatitis pain? Gastroenterology. 2013 Mar;144(3):e18. doi: 10.1053/j.gastro.2012.12.033. Epub 2013 Jan 25. No abstract available. PMID 23357056
- [Background] Dimcevski G, Sami SA, Funch-Jensen P, Le Pera D, Valeriani M, Arendt-Nielsen L, Drewes AM. Pain in chronic pancreatitis: the role of reorganization in the central nervous system. Gastroenterology. 2007 Apr;132(4):1546-56. doi: 10.1053/j.gastro.2007.01.037. Epub 2007 Jan 25. PMID 17408654
- [Background] Ceyhan GO, Demir IE, Rauch U, Bergmann F, Muller MW, Buchler MW, Friess H, Schafer KH. Pancreatic neuropathy results in "neural remodeling" and altered pancreatic innervation in chronic pancreatitis and pancreatic cancer. Am J Gastroenterol. 2009 Oct;104(10):2555-65. doi: 10.1038/ajg.2009.380. Epub 2009 Jun 30. PMID 19568227
- [Background] Nguyen-Tang T, Dumonceau JM. Endoscopic treatment in chronic pancreatitis, timing, duration and type of intervention. Best Pract Res Clin Gastroenterol. 2010 Jun;24(3):281-98. doi: 10.1016/j.bpg.2010.03.002. PMID 20510829
- [Background] Talukdar R, Murthy HV, Reddy DN. Role of methionine containing antioxidant combination in the management of pain in chronic pancreatitis: a systematic review and meta-analysis. Pancreatology. 2015 Mar-Apr;15(2):136-44. doi: 10.1016/j.pan.2015.01.003. Epub 2015 Jan 21. PMID 25648074
- [Background] Olesen SS, Bouwense SA, Wilder-Smith OH, van Goor H, Drewes AM. Pregabalin reduces pain in patients with chronic pancreatitis in a randomized, controlled trial. Gastroenterology. 2011 Aug;141(2):536-43. doi: 10.1053/j.gastro.2011.04.003. Epub 2011 Apr 14. PMID 21683078
- [Background] Bloechle C, Izbicki JR, Knoefel WT, Kuechler T, Broelsch CE. Quality of life in chronic pancreatitis--results after duodenum-preserving resection of the head of the pancreas. Pancreas. 1995 Jul;11(1):77-85. doi: 10.1097/00006676-199507000-00008. PMID 7667246
- [Background] Hallstrom H, Norrbrink C. Screening tools for neuropathic pain: can they be of use in individuals with spinal cord injury? Pain. 2011 Apr;152(4):772-779. doi: 10.1016/j.pain.2010.11.019. Epub 2011 Jan 26. PMID 21272997
- [Background] Fitzsimmons D, Kahl S, Butturini G, van Wyk M, Bornman P, Bassi C, Malfertheiner P, George SL, Johnson CD. Symptoms and quality of life in chronic pancreatitis assessed by structured interview and the EORTC QLQ-C30 and QLQ-PAN26. Am J Gastroenterol. 2005 Apr;100(4):918-26. doi: 10.1111/j.1572-0241.2005.40859.x. PMID 15784041
- [Background] • S Sarkar, D Hazarika, A Adak, P Sarkar, M Khan, NR Duvvur, R Talukdar. Impact of Personalized Counseling on Depression and Quality of Life in Patients with Chronic Pancreatitis: Results from a Randomized Controlled Trial Gastroenterology 156 (6), S-166.
- [Background] • S Sarkar, N Reddy, R Talukdar. Determinants of depression and its impact on quality of life in patients with chronic pancreatitis. Gut 67 (Suppl 2), A79-A80.